CLINICAL TRIAL: NCT01419925
Title: A Phase II Multicenter, Randomized, Placebo Controlled Study to Assess the Safety and Immunogenicity of an IM Influenza Vaccine (Multimeric-001) Followed by Administration of TIV to Elderly Volunteers.
Brief Title: A Study to Assess the Safety and Immunogenicity of M-001 Influenza Vaccine as a Primer to TIV in Elderly Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BiondVax Pharmaceuticals ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BVX-005
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Influenza; Healthy
Keywords: influenza vaccine; peptide; universal; prime; boost; TIV; HAI; Hemagglutination Inhibition; elderly
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Two Multimeric-001 administrations followed by TIV
  Interventions: Biological: Two Multimeric-001 administrations followed by TIV
- Group B (Experimental): One administration of Multimeric-001 followed by TIV
  Interventions: Biological: One administration of Multimeric-001 followed by TIV
- Group C (Experimental): One administration of adjuvanted M-001 followed by TIV
  Interventions: Biological: One administration of adjuvanted M-001 followed by TIV
- Group D (Active Comparator): One administration of placebo followed by TIV
  Interventions: Biological: One administration of placebo followed by TIV

INTERVENTIONS:
Biological: Two Multimeric-001 administrations followed by TIV — Two administrations of non adjuvanted M-001, 500 mcg followed by TIV at intervals of 19-23 days
  Arms: Group A
Biological: One administration of Multimeric-001 followed by TIV — One administration of non adjuvanted Multimeric-001, 500 mcg, followed by TIV at intervals of 19-23 days
  Arms: Group B
Biological: One administration of adjuvanted M-001 followed by TIV — One administration of adjuvanted (Aluminum phosphate) Multimeric-001, 500 mcg, followed by TIV at intervals of 19-23 days
  Arms: Group C
Biological: One administration of placebo followed by TIV — One administration of saline (Placebo)followed by TIV at intervals of 19-23 days (serving as an active comparator)
  Arms: Group D

SUMMARY:
"Multimeric-001" (M-001) has been recently developed, containing conserved, common linear influenza epitopes that activate both cellular and humoral arms of the immune system against a wide variety of influenza A and B strains. Apart from its direct action, M-001 is an attractive candidate for priming immune responses to seasonal influenza vaccine in the elderly population. The current clinical study was designed to assess M-001's standalone and priming action in subjects over 65 years old.

This is a second Phase II study comprising 120 participants. Eligible subjects were randomized to receive to receive either two sequential non-adjuvanted or a single non-adjuvanted or a single adjuvanted intramuscular injection of 500 mcg M-001 (treatment), or one placebo (saline) injection, before receiving the TIV.

DETAILED DESCRIPTION:
This was a two-center, randomized, placebo-controlled study. 120 subjects were randomized 1:1:1:1 into four groups to receive either two sequential non-adjuvanted or a single non-adjuvanted or a single adjuvanted intramuscular injection of 500 mcg M-001 (treatment), or one placebo (saline) injection, before receiving the TIV. Due to visual differences between placebo and treatment the study was partially blinded. Hemagglutinin inhibition (HAI) was evaluated at baseline and 3 weeks after standard trivalent inactivated influenza vaccine (TIV) vaccination as a measure of M-001's efficacy. Cell mediated immune (CMI) responses were also evaluated in some of the subjects who received non-adjuvanted and adjuvanted M-001 vaccinations. The subjects were monitored for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at the age of at least 65 years old
* Eligible to receive the standard seasonal influenza vaccine according to the MOH guidelines.
* Subjects who provide written informed consent to participate in the study.
* Subjects able to adhere to the visit schedule and protocol requirements and are available to complete the study.
* Haematology, chemistry and urinalysis values with no clinical significance or do not reflect a medical condition which, according to the physician's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Male subjects must agree to use a condom during the full term of the study period (including follow up) if female partner is not using an acceptable contraceptive method.
* Subjects who are seronegative to at least one of the strains included in the seasonal vaccine against influenza for 2011- 2012

Exclusion Criteria:

* Known history of significant medical disorder which, in the investigator's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Subjects with known Guillain Barré Syndrome in the past.
* Subjects who have been immunized with anti-influenza vaccine or infected by influenza virus within eight months prior to the screening visit.
* Known hypersensitivity associated with previous influenza vaccination.
* Use of an influenza antiviral medication within 4 weeks of vaccination.
* Known hypersensitivity and/or allergy to any drug or vaccine.
* Known hypersensitivity to egg proteins (eggs or egg products), chicken proteins, or any of the components of the commercial vaccine (e.g., formaldehyde, and octoxinol 9 (Triton X-100) and neomycin).
* Persons deficient in producing antibodies, whether due to genetic defect, immunodeficiency disease, or immunosuppressive therapy.
* History of any bleeding disorder or subjects with thrombocytopenia (since bleeding may occur following an intramuscular administration to these subjects).
* Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at screening visit which, according to the physician's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Positive serology for HIV, HCV antibody or HBsAg.
* Any acute medical situation (e.g. acute infection, ongoing flu symptoms) with or without fever within 48 hours of vaccination, which is considered significant by the Investigator.
* Subjects who participated in another interventional clinical study within 30 days prior to first dose
* Subjects who are non-cooperative or unwilling to sign consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 63 days
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability were similar (not statistically significant) in the experimental and control group
  Number of Participants with Adverse Events possible/probably related to the study drug in each treatment group:
  Group A: Twice M-001 - 9 AEs Group B: Once M-001 - 5 AEs Group C: Once Alum-M-001 - 13 AEs Group D: Placebo - 7 AEs

SECONDARY OUTCOMES:
Immunity induced by priming and boosting, measured by HAI | 21 days after boost immunization with TIV
  Hemagglutination Inhibition (HAI) test for anti influenza antibodies to TIV strains revealed an elevated proportion of participants achieving seroconversion in the groups primed with M-001 and boosted with TIV, as compared to participants given TIV alone. The viruses contained in the TIV were A/California/7/09, A/Perth/16/09 or B/Brisbane/60/08 . Enhanced Seroconversion and GMT post immunization were found in the experimental group primed with either adjuvanted or non adjuvanted M-001. Note that the superior HAI responses were demonstrated for both seasonal (H3N2 and B strain) and pandemic strains (swine H1N1 strain that is contained in the TIV).
Cellular immunity | 21 days after M-001 immunization
  Intracellular staining followed by FACS analysis of CD4/CD8 lymphocytes secreting IFN gamma showed elevated proportions of CD4+ cells secreting IFN gamma following exposure of PBMC from subjects immunized with M-001 to influenza antigens and to M-001. Note that the test was performed before boosting with TIV and hence demonstrates the cross immunity offered by immunization with M-001 alone and suggests a CD4+ mediated mechanism of action for M-001 as a universal primer.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jacob Atzmon, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Hadassah medical center, Jerusalem, Israel

REFERENCES:
- [Derived] Atsmon J, Caraco Y, Ziv-Sefer S, Shaikevich D, Abramov E, Volokhov I, Bruzil S, Haima KY, Gottlieb T, Ben-Yedidia T. Priming by a novel universal influenza vaccine (Multimeric-001)-a gateway for improving immune response in the elderly population. Vaccine. 2014 Oct 7;32(44):5816-23. doi: 10.1016/j.vaccine.2014.08.031. Epub 2014 Aug 28. PMID 25173483